CLINICAL TRIAL: NCT00226304
Title: The Evaluation of Focal Contrast-Enhancing Brain Lesions in HIV-Infected Patients
Brief Title: Evaluation of Brain Lesions in HIV-infected Patients for Diagnosis of Primary Central Nervous System Lymphoma
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050246; 05-CC-0246
Record Dates: First submitted 2005-09-23; First posted 2005-09-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-15

CONDITIONS: HIV Infections; Lymphoma, AIDS-Related
Keywords: Focal Brain Lesions; AIDS; Lymphoma; EBV; FDG-PET; HIV Infection; Brain Lesion
MeSH Terms: conditions — HIV Infections; Lymphoma, AIDS-Related; Acquired Immunodeficiency Syndrome; Lymphoma

SUMMARY:
This study will evaluate the usefulness of two tests in quickly distinguishing whether a patient with HIV infection and focal brain lesions (an injury in a specific area of the brain) has a rare type of cancer called primary central nervous system lymphoma (PCNSL), or a parasitic infection called toxoplasmic encephalitis.

Toxoplasmic encephalitis is caused by a parasite and can be treated with antibiotics. PCNSL (lymphoma of the brain or spinal cord) must be definitively diagnosed with a brain biopsy (removal of a small piece of brain tissue), and the treatment is radiation therapy and chemotherapy.

The tests under study for diagnosing PCNSL or toxoplasmic encephalitis are measurement of Epstein Barr virus (EBV) DNA in cerebrospinal fluid (CSF) and FDG-PET scan of the brain. EBV is often found in the CSF of people with PCNSL. The study also will compare the accuracy of two imaging techniques-TI-SPECT and FDG-PET-in distinguishing between toxoplasmosis and PCNSL.

Patients 18 years of age and older who have HIV infection and at least one focal brain lesion without a prior history of PCNSL or toxoplasmic encephalitis may be eligible for this study. Each candidate is screened with a medical history, physical examination, blood and urine tests and MRI scans of the brain.

Upon entering the study, all participants take medication to treat toxoplasmic encephalitis. They undergo lumbar puncture (spinal tap) to obtain CSF for analysis, an FDG-PET scan, and a 201TI-SPECT scan. For the PET scan, a radioactive substance is injected into an arm, followed by scanning in a doughnut-shaped machine similar to a CT scanner. SPECT is similar to PET but uses a different radioactive tracer, and the patient lies on a table while the SPECT camera rotates around the patient's head. Patients whose test results indicate a low risk for lymphoma continue antibiotic therapy for toxoplasmosis. They have repeat MRI scans around 4, 7, and 14 days after starting the drug to monitor the response to therapy. Antiretroviral therapy is initiated in patients who are not already on such a regimen.

Patients whose test results indicate a high risk for PCNSL have a CT scan to look for evidence of lymphoma elsewhere in the body and are referred for consultation with a neurosurgeon to discuss undergoing a brain biopsy. The brain biopsy is done in the operating room under general anesthesia. A small cut is made in the scalp and a small opening is made in the skull over the area of the brain to be biopsied. A needle is placed in the opening in the skull and, guided by CT or MRI, moved to the abnormal area of the brain, where a small piece of tissue is removed for study under a microscope.

Patients found to have toxoplasmosis are discharged from the hospital to the care of their primary care physician after they are getting better and are tolerating all their medications. They return to NIH for follow-up visits about 4 weeks, and 6 months after discharge.

Patients found to have lymphoma are referred to the National Cancer Institute for screening for enrollment in a treatment protocol. Patients who are not eligible for a treatment protocol are referred back to their primary care physician or for another NIH treatment protocol, if one is available. Patients with lymphoma are seen at the NIAID outpatient clinic for follow-up visits and laboratory examinations every 3 months for 2 years.

DETAILED DESCRIPTION:
Epstein Barr Virus (EBV)-associated primary central nervous system lymphoma (PCNSL) remains a major problem among AIDS patients. The clinical presentation is often clinically indistinguishable from toxoplasmic encephalitis. The method of choice for establishing the definitive diagnosis is brain biopsy. This procedure can be associated with a significant morbidity and mortality, and therefore less invasive means of diagnosing cerebral mass lesions have been studied.

Currently, an accepted standard of care for HIV-infected patients that present with signs and symptoms of focal brain lesions is to empirically treat for toxoplasmic encephalitis. Brain biopsy is often deferred until there is demonstration of lack of clinical response or progression on empiric therapy. As a result, treatment initiation is frequently delayed. During this time it is not unusual for further clinical deterioration to occur before appropriate therapies can be initiated. Frequently, the alternative approaches then become a question of appropriate palliation rather than curative intent therapy.

Less invasive diagnostic tests to assist in the diagnosis have been investigated. Based on the finding that essentially 100% of HIV-related PCNSL are EBV-associated, the detection of EBV DNA by PCR amplification in the cerebrospinal fluid (CSF) has demonstrated clinical usefulness in the diagnosis, as has the use of neuroradiologic imaging to detect the malignancy. Prior studies have demonstrated that the use of a combination of neuroradiologic, immunologic, and clinical variables in the workup of focal brain lesions in HIV-infected patients to be quite accurate in identifying patients in need of brain biopsy, but a diagnostic algorithm that incorporates the combination of the most sensitive and specific tests in a timely manner has not yet been explored.

This study seeks to evaluate an algorithm for the workup of HIV infected patients with focal brain lesions so as to expedite the diagnosis and subsequent treatment of PCNSL. The goals of the study are to 1) determine the specificity, sensitivity, and positive predictive value of a diagnostic algorithm that entails the use of the combination of EBV detection in the CSF and FDG-PET scanning to diagnose PCNSL; 2) evaluate the time to response to anti-toxoplasmic encephalitis therapy, and 3) evaluate the sensitivities and specificities of FDG-PET and (201)Tl-SPECT scanning in identifying PCNSL. Up to one hundred HIV-infected patients with history of at least one focal brain lesion will be screened for enrollment. All patients will be treated empirically for toxoplasmic encephalitis until an alternative diagnosis is confirmed. All enrolled patients will be treated concurrently with antiretroviral therapy. Patients identified to have PCNSL will be referred to the NCI Treatment of PCNSL Protocol for further treatment if the study is open for enrollment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adult (18 years old or older) HIV-infected patient

HIV infected by OraQuick rapid test using saliva, venipuncture whole blood, or fingerstick whole blood; or by reactive ELISA and Western Blot as determined by an outside CLIA-approved laboratory facility or by NIH Clinical Pathology Laboratory or SAIC-Frederick Inc Monitoring Laboratory. HIV infection as determined by an outside CLIA-approved laboratory facility will be verified by a standard HIV-1 ELISA with Western Blot confirmation prior to brain biopsy.

Evidence of contrast-enhancing focal brain lesion(s) as seen on MRI or CT

Willingness to give informed consent and provided by Durable Power of Attorney. In the event that no Durable Power of Attorney has been designated and the patient is unable to do so, the NIH Ethics Committee will be consulted. All patients must designate a Durable Power of Attorney in order to participate in the study.

Willingness to undergo the procedures involved in the diagnostic evaluation: lumbar puncture, FDG-PET scan, 201Tl-SPECT scan, and brain biopsy.

Permit the storage of blood, CSF, and tissue samples for future research use

Willingness to undergo HLA testing

EXCLUSION CRITERIA:

Previous PCNSL

History of prior malignancy other than PCNSL unless in remission for 1 year or longer; non-melanoma skin cancer and Kaposi's sarcoma excepted

History of previous diagnosis of toxoplasmic encephalitis or other CNS infection causing focal contrast-enhancing brain lesions

Pregnancy or currently breast feeding

Have any other condition that the research team considers a contraindication to participating in the study, e.g. severe cardiac, renal, or pulmonary dysfunction.

Weight greater than 400 lb for PET and 500 lb for SPECT (limit of the gantry).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-09-20; Study Completion 2009-04-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cote TR, Manns A, Hardy CR, Yellin FJ, Hartge P. Epidemiology of brain lymphoma among people with or without acquired immunodeficiency syndrome. AIDS/Cancer Study Group. J Natl Cancer Inst. 1996 May 15;88(10):675-9. doi: 10.1093/jnci/88.10.675. PMID 8627644
- [Background] Basso U, Brandes AA. Diagnostic advances and new trends for the treatment of primary central nervous system lymphoma. Eur J Cancer. 2002 Jul;38(10):1298-312. doi: 10.1016/s0959-8049(02)00031-x. PMID 12091059
- [Background] MacMahon EM, Glass JD, Hayward SD, Mann RB, Becker PS, Charache P, McArthur JC, Ambinder RF. Epstein-Barr virus in AIDS-related primary central nervous system lymphoma. Lancet. 1991 Oct 19;338(8773):969-73. doi: 10.1016/0140-6736(91)91837-k. PMID 1681341